CLINICAL TRIAL: NCT06073301
Title: Comparison of Treatment with Acellular Fish Skin (AFS) to Acellular Human Cadaver Allograft (AHC) in the Treatment of Necrotizing Fasciitis (NF)
Brief Title: AFS Compared to AHC in Treatment of Necrotizing Fasciitis NF
Acronym: NF
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Kerecis Ltd. (Industry)
Collaborators: Joseph M. Still Research Foundation, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KS-0820
Record Dates: First submitted 2023-09-21; First posted 2023-10-10 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-10

CONDITIONS: Necrotizing Fasciitis
MeSH Terms: conditions — Fasciitis, Necrotizing

STUDY DESIGN:
Intervention Model Description: Eligible Subjects for this single center open label randomized study, will randomize eligible subjects to 2 groups, 15 in the treatment arm (Fish skin graft) and 15 in the control arm (cadaver graft). Randomization will be done electronically on day of surgery, enrollment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Treatment: Acellular Fish Skin (AFS) with Standard of Care Negative Pressure Wound Therapy (NPWT) (Experimental): Eligible subjects will be randomized electronically to either the Acellular Fish Skin (AFS)arm. The subject will undergo wound bed preparation by surgical debridement. the AFS will be applied to the wound bed and secured with sutures, the size of the AFS will be determined after surgical debridement. Once the AFS is in place a Negative Pressure Wound Therapy device will be placed. the subject will be monitored weekly on scheduled intervals of +/- 4 days post AFS placement to assess the status of the wound and readiness for autografting. Once the wound is ready for autografting the subject will be monitored for autograft take, for up to 9 visits. Long term follow-up will be done at month 3, 6, 9 post autograft placement
  Interventions: Device: Acellular Fish Skin Graft (AFS) with Standard of Care Negative Pressure Wound Therapy (NPWT)
- Acellular Human Cadaver with Standard of Care Negative Pressure Wound Therapy (NPWT) (Active Comparator): .Eligible subjects will be randomized electronically to standard of care arm which is Acellular Human Cadaver (AHC) The subject will undergo wound bed preparation by surgical debridement. The AHC will be applied to the wound bed and secured with sutures, the size of the AHC will be determined after surgical debridement. Once the AHC is in place a Negative Pressure Wound Therapy device will be placed. the subject will be monitored weekly on scheduled intervals of +/- 4 days post AHC placement to assess the status of the wound and readiness for autografting. Once the wound is ready for autografting the subject will be monitored for autograft take, for up to 9 visits. Long term follow-up will be done at month 3, 6, 9 post autograft placement
  Interventions: Other: Acellular Human Cadaver (AHC) with Standard of care Negative Pressure Wound Therapy (NPWT)

INTERVENTIONS:
Device: Acellular Fish Skin Graft (AFS) with Standard of Care Negative Pressure Wound Therapy (NPWT) — Acellular Fish Skin, used to temporize a wound bed prior to autograft. The intention is to prepare the wound bed for optimal autograft take.
  Other Names: Brand Kerecis: GraftGuide, GraftGuide Micro, GraftGuide Meshed
  Arms: Treatment: Acellular Fish Skin (AFS) with Standard of Care Negative Pressure Wound Therapy (NPWT)
Other: Acellular Human Cadaver (AHC) with Standard of care Negative Pressure Wound Therapy (NPWT) — Acellular Human Cadaver , used to temporize a wound bed prior to autograft. The intention is to prepare the wound bed for optimal autograft take.
  Other Names: AHC
  Arms: Acellular Human Cadaver with Standard of Care Negative Pressure Wound Therapy (NPWT)

SUMMARY:
Necrotizing Fasciitis (NF) is a potentially life-threatening soft tissue infection. This study is comparing acellular fish skin graft (AFS) to standard of care allograft (AHC) in the treatment of NF. The purpose of this study is to compare clinical outcomes and time until autograft take in patients that were treated with AHC or AFS prior to permanent autografting to treat NF.

DETAILED DESCRIPTION:
This will be a prospective, randomized, open-label, interventional, single-center study looking at time to autograft placement and time to full closure in subjects treated with acellular fish skin compared to subjects treated with acellular human cadaver skin to prepare the wound bed prior to grafting. Subjects eligible to receive study treatment will be any adult patient (18 years of age or older) admitted to the Joseph M. Still Burn Center or Advanced Wound Clinic at Doctors Hospital Augusta with a diagnosis of NF that has been treated and is stable. Prior wound excisions will be allowed until the surgeon has deemed the wound stable and free from necrotizing processes.

Exclusion criteria will be positive pregnancy test on admission, subject has active diagnosis of any autoimmune process, or cancer that in the opinion of the investigator would prevent the subject from successfully participating in the study.

ELIGIBILITY:
Inclusion Criteria:

* Is ≥18 years of age.
* Has been admitted to the Joseph M. Still Burn Center at Doctors Hospital Augusta or Advanced Wound Clinic for treatment of NF which has been treated and is considered stable.

Exclusion Criteria:

* Subject has been previously enrolled into this study or is currently participating in another drug or device study that has not reached its primary endpoint.
* Index wounds that due to anatomical location are unable to apply a NPWT device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint: To compare the time from first application of study product to time of autografting between the two study groups. | 9 weeks
  To compare the time (number of days) from the first application of study product to time (number of days ) to autografting.

SECONDARY OUTCOMES:
Secondary Endpoint: To compare the percentage of autograft take between the two study groups. | 9 weeks
  To measure the percentage from 0 to 100% of autograft adherence to the wound bed

CONTACTS AND LOCATIONS:
Overall Officials: Bounthavy Homsombath, MD, Principal Investigator — Joseph M.Still Research Foundation
Locations (1):
- Joseph M. Still Research Foundation, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No